CLINICAL TRIAL: NCT04690049
Title: An Innovative Therapeutic Exercise Approach Based on Load Progression Criteria for the Management of Shoulder Impingement Syndrome: a Randomized Controlled Trial
Brief Title: Therapeutic Progressive Exercise on Shoulder Impingement Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Antonio I Cuesta-Vargas, Professor, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ProgEx-01
Record Dates: First submitted 2020-12-21; First posted 2020-12-30 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-09

CONDITIONS: Shoulder Impingement; Tendinopathy
Keywords: shoulder impingement syndrome; tendinopathy; exercise
MeSH Terms: conditions — Shoulder Impingement Syndrome; Tendinopathy; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular resistance exercise group (Experimental): Subjects will develop an innovator program consisting in the performance of exercises of increasing difficulty, with movements based on functional tests to analyze the subjects' neuromuscular capacities. Participants will attend to 80 individual, face-to-face physiotherapy sessions, including both supervised and semi-supervised monitoring. From the total, a minimum of 15 sessions will be supervised, including 6 sessions to teach and monitor the exercises, and 9 sessions to perform the tests in order to quantify the load; 37 sessions will be semi-supervised, where subjects will perform the exercises independently, but with the presence of an instructor; additionally, the remaining 28 sessions will consist in non-supervised aerobic work at a 70-80% from maximum heart rate, obtained according to the methodology of Tanaka et al.
  Interventions: Other: Neuromuscular resistance exercise program
- Control exercise group (Active Comparator): This program will be based on a home exercise protocol considering painful sensation and self-perceived stability as progression criteria: regarding pain management, exercises will be planned in a way that increased pain after their performance reverts to before-exercise levels prior to the next session; regarding self-perceived stability, participants will be asked to maintain a constant sensation of joint stability and control during the execution of the exercises. Participants will perform shoulder rotations (external and internal) and abduction up to 30º by using elastic bands. The resistance of the band will be adjusted by the physiotherapist so that participants perceive the exercises as demanding enough but not too unpleasant, being able to complete the 10 repetitions before taking the rest. Likewise, exercises will progress until a maximum of 90º of shoulder abduction.
  Interventions: Other: Control exercise program with elastic band

INTERVENTIONS:
Other: Neuromuscular resistance exercise program — This neuromuscular resistance exercise program will be organized in 5 stages, distributing the different phases in 2, 4, 4, 2 and 2 weeks respectively, with a frequency of 3 sessions/week. In addition, 2 weekly sessions of aerobic work with cycloergometer will be developed. The duration of each session will last 30 minutes. The parameters of load and execution speed will be modified as the exercise program progresses along the phases, with the goal of have an impact on the different aspects of the neuromuscular system.
  Arms: Neuromuscular resistance exercise group
Other: Control exercise program with elastic band — This program is based on previous literature so that it remains comparable to the experimental program.
  The parameters will consist in 3 sets of 10 repetitions, 2 times/day, 3 times/week, for a total of 6 weeks.
  Arms: Control exercise group

SUMMARY:
Upper limb tendinopathies, especially the so called "shoulder impingement syndrome", is a common injury among the population. Its management usually involves active treatments, being the therapeutic progressive exercise the most important and effective modality. However, whether a certain criterion is more appropriate than another when progressing the exercise program remains unclear. We propose a new program based on progressive exercises serving as a standard approach for the management of shoulder impingement syndrome.

DETAILED DESCRIPTION:
Shoulder pain is a common condition affecting our society. It is estimated that between 7 and 67% of the adult population will suffer from shoulder pain at least once in their lifetime. Some research suggest that shoulder impingement syndrome (SIS) is responsible for 44 to 60% from the medical consultations regarding shoulder pain with an approximate prevalence of 70-200 per 1000 adults, which implies a remarkable use of health care resources.

Among all the musculoskeletal injuries affecting the shoulder complex, SIS remains as the most common condition, characterized for leading to loss function and disability. Its pathogenesis is associated with the affection of diverse structures and tissues like the subacromial bursa, rotator cuff tendons, acromion, coracoacromial ligament and the long head of biceps brachii. The etiology of this condition comprises multiple causes, including capsular tightness, alteration of shoulder kinematics with scapula dysfunction and muscle imbalance, and also the overuse factor.

Treatment modalities to deal with SIS embrace both surgical procedures, i.e., arthroscopic subacromial decompression) and conservative approaches (i.e., physical therapy), becoming the therapeutic exercise increasingly popular due to arising evidence from the last 30 years. Furthermore, with regard to potential effects, therapeutic exercise presents itself as a safer and less aggressive alternative, causing fewer adverse effects than pharmacological or surgical options, which are relegated preferably as secondary choices.

There is a wide evidence supporting the exercise therapy as an effective strategy for the management of SIS. However, some controversy exists regarding the optimal approach in terms of intensity, frequency and number of repetitions. Thus, a program acting as a gold standard for the development and progression of the proposed exercises is still lacking, especially when attempting to estimate the pure effect of progressive exercise in isolation between experimental and control group.

Prior research evaluating the effect of progressive exercise for the management of SIS usually included programs with a duration of 3 months. However, other studies established follow-up periods of either one month and a half or, conversely, more than 6 months. That, together with the wide variety of post-treatment follow-ups, makes it difficult to find the optimal period where the results derived inherently from the intervention and not from the natural course of the condition may be observed.

Regarding the progression criteria, there seems to be a tendency to consider the modulation of the painful sensation as the main benchmark from which the exercise may progress in difficulty, but some other progression sub-criteria can also be found, such as fatigue or subjective perception. Furthermore, the presence of other conditioning elements, like proximity to pain threshold or a certain reference value in the Visual Analogue Scale (VAS), reduces the homogeneity among the exercise programs and hinders the standardization of the ideal exercise progression when performing the exercises for the management of SIS.

The main objective of this clinical trial is to prove the efficacy of a progressive exercise program based on strength and resistance training in comparison to an exercise protocol from the literature to increase neuromuscular and cardiorespiratory capacities and improve the symptoms in subjects with SIS. In addition, we propose to determine the existence or not of statistically significant differences between treatment modalities by evaluating whether these changes occur before, during or after the application of the proposed exercise protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subjects older than 18 years.
* Subjects previously diagnosed with shoulder impingement syndrome.
* Presence of 3 of the following sings: impingement sign according to Neer and to Hawking-Kennedy, positive result on Jobes test, painful arc, and positive result on Patte's manoeuvre.

Exclusion Criteria:

* Findings of spinal radiculopathy.
* General neck and shoulder pain.
* Symptoms of frozen shoulder.
* Pregnancy.
* Fybromyalgia.
* Suspected polyarthritis.
* Chronic pain syndrome.
* Altered blood coagulation.
* Consumption of anticoagulants, opioids or antiepileptics.
* Drug intakes.
* Alcohol intakes higher than 27.4 grams for men or 13.7 grams for women.
* Allergies.
* Cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Function measured with Disability of the Arm, Shoulder and Hand (DASH) | 14 weeks
  Functional scores from Disability of the Arm, Shoulder and Hand (DASH) questionnaire.
  Score ranges from 0 (no disability) to 100 (most severe disability)
Change from baseline in Function measured with Constant-Murley Score (CMS) | 14 weeks
  Functional scores from Constant-Murley Score (CMS) Constant-Murley score (CMS) is a 100-points scale: the higher the score, the higher the quality of the function.
Change from baseline in Function measured with Upper Limb Functional Index (ULFI) | 14 weeks
  Functional scores from Upper Limb Functional Index (ULFI) Score ranges from 0 (no disability) to 25 (most severe disability)
Change from baseline Painful Sensation | 14 weeks
  Pain scores from Visual Analogue Scale (VAS) Score ranges from 0 (no pain) to 10 (most severe pain)
Change from baseline Range of motion (ROM) | 14 weeks
  Active shoulder joint ROM (flexion, extension, abduction, internal/external rotations) by goniometry
Change from baseline Subacromial Space | 14 weeks
  Measurement of subacromial space by ultrasonography

SECONDARY OUTCOMES:
Change from baseline Quality of Life | 14 weeks
  Quality of life scores from EuroQol-5D questionnaire
  EQ-5D embodies two components:
  * Health state description: subjects select one of three different levels of problem severity within each of five health domains. The levels are none, moderate and severe/extreme (coded 1 through 3, respectively), whilst the domains are mobility, capacity for self-care, conduct of usual activities, pain/discomfort and anxiety/depression.
  * Evaluation: using a visual analogue scale (VAS), ranging from 0 ("worst imaginable health state") and at 100 ("best imaginable health state")
Change from baseline Health Status | 14 weeks
  Health status scores from Short-Form 12 (SF-12) questionnaire SF-12 gathers information from eight domains: the higher the scores, the better the health)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Cuesta-Vargas, PhD, Study Chair — University of Malaga

IPD SHARING:
Plan to Share IPD: Undecided
If further decided, IPD will be shared under request.

REFERENCES:
- [Background] Luime JJ, Koes BW, Hendriksen IJ, Burdorf A, Verhagen AP, Miedema HS, Verhaar JA. Prevalence and incidence of shoulder pain in the general population; a systematic review. Scand J Rheumatol. 2004;33(2):73-81. doi: 10.1080/03009740310004667. PMID 15163107
- [Background] Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Phys Ther. 2000 Mar;80(3):276-91. PMID 10696154
- [Background] Marin-Gomez M, Navarro-Collado MJ, Peiro S, Trenor-Gomis C, Paya-Rubio A, Bernal-Delgado E, Hernandez-Royo A. [The quality of care in shoulder pain. A medical audit]. Gac Sanit. 2006 Mar-Apr;20(2):116-23. doi: 10.1157/13087322. Spanish. PMID 16753088
- [Background] Kuhn JE. Exercise in the treatment of rotator cuff impingement: a systematic review and a synthesized evidence-based rehabilitation protocol. J Shoulder Elbow Surg. 2009 Jan-Feb;18(1):138-60. doi: 10.1016/j.jse.2008.06.004. Epub 2008 Oct 2. PMID 18835532
- [Background] Seitz AL, McClure PW, Finucane S, Boardman ND 3rd, Michener LA. Mechanisms of rotator cuff tendinopathy: intrinsic, extrinsic, or both? Clin Biomech (Bristol). 2011 Jan;26(1):1-12. doi: 10.1016/j.clinbiomech.2010.08.001. Epub 2010 Sep 16. PMID 20846766
- [Background] Cardoso TB, Pizzari T, Kinsella R, Hope D, Cook JL. Current trends in tendinopathy management. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):122-140. doi: 10.1016/j.berh.2019.02.001. Epub 2019 Mar 8. PMID 31431267
- [Background] Cook JL. Ten treatments to avoid in patients with lower limb tendon pain. Br J Sports Med. 2018 Jul;52(14):882. doi: 10.1136/bjsports-2018-099045. Epub 2018 Feb 23. No abstract available. PMID 29475840
- [Background] Hallgren HC, Holmgren T, Oberg B, Johansson K, Adolfsson LE. A specific exercise strategy reduced the need for surgery in subacromial pain patients. Br J Sports Med. 2014 Oct;48(19):1431-6. doi: 10.1136/bjsports-2013-093233. Epub 2014 Jun 26. PMID 24970843
- [Background] Holmgren T, Oberg B, Sjoberg I, Johansson K. Supervised strengthening exercises versus home-based movement exercises after arthroscopic acromioplasty: a randomized clinical trial. J Rehabil Med. 2012 Jan;44(1):12-8. doi: 10.2340/16501977-0889. PMID 22124602
- [Background] Osteras H, Torstensen TA, Osteras B. High-dosage medical exercise therapy in patients with long-term subacromial shoulder pain: a randomized controlled trial. Physiother Res Int. 2010 Dec;15(4):232-42. doi: 10.1002/pri.468. PMID 21110409
- [Background] Brox JI, Gjengedal E, Uppheim G, Bohmer AS, Brevik JI, Ljunggren AE, Staff PH. Arthroscopic surgery versus supervised exercises in patients with rotator cuff disease (stage II impingement syndrome): a prospective, randomized, controlled study in 125 patients with a 2 1/2-year follow-up. J Shoulder Elbow Surg. 1999 Mar-Apr;8(2):102-11. doi: 10.1016/s1058-2746(99)90001-0. PMID 10226960
- [Background] Ketola S, Lehtinen JT, Arnala I. Arthroscopic decompression not recommended in the treatment of rotator cuff tendinopathy: a final review of a randomised controlled trial at a minimum follow-up of ten years. Bone Joint J. 2017 Jun;99-B(6):799-805. doi: 10.1302/0301-620X.99B6.BJJ-2016-0569.R1. PMID 28566400
- [Background] Heron SR, Woby SR, Thompson DP. Comparison of three types of exercise in the treatment of rotator cuff tendinopathy/shoulder impingement syndrome: A randomized controlled trial. Physiotherapy. 2017 Jun;103(2):167-173. doi: 10.1016/j.physio.2016.09.001. Epub 2016 Sep 21. PMID 27884499
- [Background] Tyler TF, Nicholas SJ, Roy T, Gleim GW. Quantification of posterior capsule tightness and motion loss in patients with shoulder impingement. Am J Sports Med. 2000 Sep-Oct;28(5):668-73. doi: 10.1177/03635465000280050801. PMID 11032222
- [Background] Miranda H, Viikari-Juntura E, Martikainen R, Takala EP, Riihimaki H. A prospective study of work related factors and physical exercise as predictors of shoulder pain. Occup Environ Med. 2001 Aug;58(8):528-34. doi: 10.1136/oem.58.8.528. PMID 11452048